CLINICAL TRIAL: NCT06745336
Title: Clinical Study of CS-001 As a Treatment for Canities (Grey Hair)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Complex Science (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS-001
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Canities; Grey Hair

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CS-001 (Experimental): CS-001 Topical Treatment
  Interventions: Drug: CS-001
- Placebo (Placebo Comparator): Placebo Topical Treatment
  Interventions: Drug: Placebo Topical Solution

INTERVENTIONS:
Drug: CS-001 — CS-001 Topical Treatment
  Arms: CS-001
Drug: Placebo Topical Solution — Placebo Topical Solution
  Arms: Placebo

SUMMARY:
Clinical Study to Assess the Safety and Efficacy of CS-001 as a treatment for Canities (Grey Hair)

DETAILED DESCRIPTION:
CS-001 is a small molecule that affects lysosomal storage and transfer of melanin from hair follicle melanocytes. In vitro and a small pilot study demonstrated re-pigmentation of grey hair following CS-001 application. The aim of this study is to assess the safety and efficacy of CS-001 as a treatment for grey hair.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 65
* Diagnosed with Grey Hair (Canities)
* Willing and able to apply the treatment as directed, comply with study
* Otherwise healthy
* Able to give informed consent

Exclusion Criteria:

* A medical history that may interfere with study objectives
* Women who are pregnant, lactating, or planning to become pregnant during the study period
* Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc)
* Subjects who have known allergies to any excipient in CS-001
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device in the treatment area within 30 days prior to study treatment initiation
* Subjects who have used any topical prescription medications in the treatment area within 30 days prior to study treatment initiation
* Subjects who have had a dermatological procedure such as surgery in the treatment area within 30 days prior to study treatment initiation
* Subject is unable to provide consent or make the allotted clinical visits

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Greying Severity Score | Week [0,52]
  Greying Severity Score (GSS). Mild Greying score between 0-5, Moderate Greying score between 6-10 and Severe Greying score between 11-15

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singal A, Daulatabad D, Grover C. Graying severity score: A useful tool for evaluation of premature canities. Indian Dermatol Online J. 2016 May-Jun;7(3):164-7. doi: 10.4103/2229-5178.182372. PMID 27294049